CLINICAL TRIAL: NCT01152970
Title: Substance Use Among Violently Injured Youth in Urban ER: Services & Outcomes
Brief Title: F.Y.I.: Flint Youth Injury Study
Acronym: FYI
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rebecca Cunningham, Professor, University of Michigan
Other Study IDs: DA024646 01A2; R01DA024646-01A2 (NIH)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Drug Usage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- drug-using youth with violent injury: Youth(ages 14-24) who report illicit drug use and who present to an urban ED for an acute violent injury
- drug-using youth with non-violent injury: Youth(ages 14-24) who report illicit drug use and who present to an urban ED for non-violence related care

SUMMARY:
The provision of medical services in an inner city Emergency Department (ED) provides a critical opportunity to identify and characterize future timing and pattern of service use among youth with drug use, who may be missed in school-based samples, and who may not yet be in the criminal justice system. Currently, there is a paucity of data on the timing, pattern, barriers, and trajectory of youth with multiple risks (illicit drug use and ED visit for acute violence related injury) in terms of their intersection with health services (substance use treatment, mental health, medical) and criminal justice system, which limits the development of optimal timing and setting for interventions. Youth treated in the ED may have exacerbated rates of illicit drug use, and other risk behaviors (i.e. delinquency, HIV risk behaviors, weapon carriage) and different trajectories of outcomes and interactions with service use sectors based on presentation for intentional injury as compared to other complaints (medical, unintentional injuries). Understanding the outcomes and service utilization among inner-city youth with drug use with and without acute violent injury is critically important in developing prevention and treatment services to address these multiple risk factors. The investigators propose a prospective observational study over a two-year period to identify a high risk group of youth with past year illicit drug use (N=650) seeking care in an inner city ED. The specific aims of the study, chosen to obtain data necessary to determine the location and content of subsequent interventions, are: (1) To describe characteristics of youth (ages 14-24; n=650) who report illicit drug use presenting to an urban ED for an acute violent injury (n=350), compared to youth with drug use who seek non-violence related ED care (n=300), including demographic characteristics, problem severity (e.g., substance use, violence, HIV risk behaviors, etc.), enabling factors, and service utilization (i.e., substance use treatment, mental health, and medical); (2) To identify the trajectories of participants' interactions with health services during the two years following their ED visit and the key characteristics (i.e., predisposing, enabling, and need factors) associated with types of service use (substance abuse treatment, mental health, and medical/ ED) and barriers to these services; and, (3) To measure two-year outcomes for this cohort and to identify key demographic and clinical characteristics of youth with drug use, who have poor outcomes in the two years after ED visit for intentional injury and other medical care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for screening:

1. youth (ages 14-24) presenting to the Hurley Medical Center (HMC) ED who are medically stable. Patients classified by medical staff as having unstable vital signs or "Level 1" trauma (e.g., unconscious, in need of immediate lifesaving procedures such as surgery), will be approached during their inpatient stay after stabilization (4% based on prior work);
2. access to a parent or guardian for consent among adolescents ages 14-17 (over 90% based on our prior work).

Positive substance use screen criteria: Youth will be eligible for the longitudinal study if they endorse on self-report computer survey past year use of illicit drugs (e.g. marijuana, cocaine, inhalants, non-prescribed use of psychoactive prescription drugs, etc).-

Exclusion Criteria:

1. youth who do not understand English
2. youth deemed unable to provide informed assent/consent by ED or research staff
3. prisoners at time of ED presentation.
4. youth who present to the ED as victims of sexual abuse or child abuse -

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients ages 14-24 seeking treatment at the Hurley Medical Center (HMC) Emergency Department (ED) located in Flint, MI will be recruited for this study.
Sampling Method: Probability Sample
Enrollment: 638 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
substance use as assessed with both the Mini-International Neuropsychiatric Interview | Change from baseline substance use at 24 month
substance use as assessed with the National Institute on Drug Abuse- Modified Alcohol, Smoking and Substance Involvement Screening Test | Change from baseline substance use at 24 month
violence behaviors as assessed with the modified Conflict Tactic Scale | Change from baseline violence behaviors at 24 month
HIV risk behaviors as assessed with the Risk Assessment Battery | Change from baseline HIV risk behaviors at 24 month
trajectories of participants' interactions with health services during the two years following their ED visit for an acute violent injury or for non-violence related care | through the study completion, over 24 months
  Services will include substance abuse treatment, mental health services, and medical services including ED recidivism and HIV testing as assessed through chart review

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Cunningham, MD, Principal Investigator — University of Michigan
Locations (1):
- Hurley Medical Center Emergency Department, Flint, Michigan, United States

REFERENCES:
- [Derived] Carter PM, Dora-Laskey AD, Goldstick JE, Heinze JE, Walton MA, Zimmerman MA, Roche JS, Cunningham RM. Arrests Among High-Risk Youth Following Emergency Department Treatment for an Assault Injury. Am J Prev Med. 2018 Dec;55(6):812-821. doi: 10.1016/j.amepre.2018.07.003. Epub 2018 Oct 19. PMID 30344036
- [Derived] Carter PM, Walton MA, Roehler DR, Goldstick J, Zimmerman MA, Blow FC, Cunningham RM. Firearm violence among high-risk emergency department youth after an assault injury. Pediatrics. 2015 May;135(5):805-15. doi: 10.1542/peds.2014-3572. Epub 2015 Apr 6. PMID 25847808
- [Derived] Cunningham RM, Ranney M, Newton M, Woodhull W, Zimmerman M, Walton MA. Characteristics of youth seeking emergency care for assault injuries. Pediatrics. 2014 Jan;133(1):e96-105. doi: 10.1542/peds.2013-1864. Epub 2013 Dec 9. PMID 24323994